

## **CONCUR – CON**tractility: **C**uff versus **UR**odynamics testing in males with voiding lower urinary tract symptoms

| Partici | Number: 8598<br>pant Identification Num | ber: | |
|---|---|---|---|
| Name of Researcher: Please <u>initial</u> | | | Please <u>initial</u> box |
| 1. | I confirm that I have read and understood the Patient Information Sheet dated 24/04/2018 (v1.0) for this study and have had the opportunity to ask questions. | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without being required to give a reason, and that this will not affect the standard of my medical care or legal rights. | | |
| 3. | I understand that relevant sections of my paper or electronic patient records may be reviewed by individuals from the research group and representatives from the Sponsor and Regulatory bodies for the purpose of audit. I give my permission for these individuals to have access to my records. | | |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | | |
| 5. | I consent to the use of ionising radiation during this study. I have read the information provided about this in the information leaflet and understand this is additional to that required for my standard test. | | |
| 6. | | | |
| Name of patient | | Signature | Date |
| Name o | f nerson receiving consent | Signaturo | Nate |

When completed: 1 for participant; 1 for medical notes; 1 (original) for researcher site file.

IRAS 231323 Page 1 of 1